CLINICAL TRIAL: NCT04534621
Title: How Brazilian Chiropractors Are Being Affected and What Strategies They Have Developed for Facing the COVID-19 Pandemic
Brief Title: How Brazilian Chiropractors Are Facing the COVID-19 Pandemic
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Trate - Tratamentos Especializados (Other)
Responsible Party: Principal Investigator, Marcelo Borges Botelho, CEO, Trate - Tratamentos Especializados
Other Study IDs: TrateTE
Record Dates: First submitted 2020-08-25; First posted 2020-09-01 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Covid19
Keywords: chiropractors; strategies; coronavirus; pandemic
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Brazilian chiropractors: A cross-sectional survey will be performed with this population (Brazilian chiropractors) to assess outcomes regarding what is the current impact and what measures they have implemented while facing the COVID-19 pandemic.
  Interventions: Other: Electronic survey

INTERVENTIONS:
Other: Electronic survey — Brazilian chiropractors will be invited by email and social media to answer an electronic survey.

SUMMARY:
Brazil has the Latin America's largest coronavirus outbreak, numbers second only to the United States in the western hemisphere. The first COVID-19 confirmed case in Brazil was on February of 2020. A 61yrs old man tested positive after returning from a trip to Italy. Few other very first cases were also imported from Europe by returning travelers. The first locally transmitted case was registered on March of 2020, when a total of 8 cases have already been confirmed. At the time the WHO declares the outbreak as a pandemic (March 11) Brazil had 52 confirmed cases being 6 of those locally transmitted.

Healthcare professionals are now more important than ever. Given the intrinsic nature of the hands-on treatment of the Chiropractic profession, it is extremely important to understand what strategies chiropractors have put in place to address patient care, safety, and self report COVID contamination of those professionals.

ELIGIBILITY:
Inclusion Criteria:

* Chiropractors graduated from national or international accredited colleges.

Exclusion Criteria:

* Chiropractors who did not treated patients in 2020.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All chiropractors from the Brazilian Chiropractic association database / thru social media / principal investigator database will be invited to participate.
Sampling Method: Non-Probability Sample
Enrollment: 948 (Estimated)
Dates: Start 2020-08-26 (Estimated); Primary Completion 2020-09-06 (Estimated); Study Completion 2020-09-18 (Estimated)

PRIMARY OUTCOMES:
What measures have been implemented to avoid SARS-COV2 transmission when taking care of patients, during the COVID-19 pandemic. | 2 weeks
  Subjects will answer a online survey addressing what measures they have implemented to prevent SARS-COV2 contamination among staff and patients, when taking care of patients. These questions address the use of individual protection devices, sanitizing methods, social distancing, patient orientation, and consultation time. These will be analyzed in conjunct, using descriptive statistics.

SECONDARY OUTCOMES:
Professionals SARS-COV2 infection rates. | 2 weeks
  Self declared SARS-COV2 infection rates.
Professional financial impact. | 2 weeks
  To assess the potential professional financial impact caused by the pandemic, the subjects will answer a question in the survey addressing if they have had a financial loss during the pandemic. This question will have the following answer options: no financial loss, less than 25% financial loss, between 25-50%, between 50-75%, more than 75% of financial loss due the pandemic.

CONTACTS AND LOCATIONS:
Overall Officials: MARCELO B BOTELHO, DC, MD, MSc, Principal Investigator — Trate

IPD SHARING:
Plan to Share IPD: No
Collective / group data sharing only.